CLINICAL TRIAL: NCT01584024
Title: Radiographic Progression of Early Caries Lesions After Resin Infiltration
Brief Title: Resin Infiltration to Arrest Early Tooth Decay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Principal Investigator, Mathilde Peters, DMD, PhD, Professor Emerita, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N010508-S3; 12-PAF02598 (Other: U-Michigan)
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Dental Caries
Keywords: Dental caries; Proximal surfaces; Posterior teeth; Carious lesions; Tooth diseases; Preventive therapy
MeSH Terms: conditions — Dental Caries; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin infiltration (Active Comparator): Resin infiltration of early caries lesion in addition to preventative measures (oral hygiene, diet counseling, repeated fluoride varnish application)
  Interventions: Device: Resin infiltration
- Control (Sham Comparator): Sham treatment of early caries lesion in addition to preventative measures (oral hygiene, diet counseling, repeated fluoride varnish application)
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Resin infiltration — Baseline treatment of one caries lesion with resin infiltration therapy, in addition to preventative measures and behavioral modification.
  ICON product: FDA-510(k): K100062
  Other Names: ICON Infiltration kit (DMG, Germany) (ICON=product name)
  Arms: Resin infiltration
Device: Sham treatment — Baseline treatment of one caries lesion with sham treatment, in addition to preventative measures and behavioral modification.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether lesion infiltration is an effective management strategy to arrest early tooth decay.

DETAILED DESCRIPTION:
A 3-year prospective, randomized control clinical trial (RCT) is designed incorporating a split mouth intra-oral design. Young volunteers (18-24 years old) with at least two early lesions in posterior teeth will be enrolled into this clinical trial to evaluate the clinical effectiveness of arresting lesion progression by resin infiltration therapy as adjunct to standard-of-care preventative measures. Lesion status (non-cavitated) is clinically confirmed prior to implementing the assigned therapy.

ELIGIBILITY:
Inclusion Criteria:

* DMFT ≥ 3 (DMFT = index of decayed-missing-filled permanent teeth)
* Having at least two early caries lesions in approximal posterior tooth surfaces
* Lesions visible on radiograph

Exclusion Criteria:

* Current participation in another clinical study
* Medically compromised subjects
* Hyposalivation
* Pregnancy
* Allergic to methylmethacrylates
* Allergic to latex
* Symptomatic teeth

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde C Peters, DMD, PhD, Study Chair — University of Michigan
Locations (1):
- Saunders USADC, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peters MC, Hopkins AR Jr, Zhu L, Yu Q. Efficacy of Proximal Resin Infiltration on Caries Inhibition: Results from a 3-Year Randomized Controlled Clinical Trial. J Dent Res. 2019 Dec;98(13):1497-1502. doi: 10.1177/0022034519876853. Epub 2019 Sep 16. PMID 31526071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caries-active volunteer cadet-candidates and cadets, at high risk for caries disease, were recruited at United States Military Academy in West-Point, New York (USA).
Pre-assignment Details: Paired, split-mouth study design: Each patient received 2 paired treatments (one of each arm). Eligible tooth pairs were selected for similarity. Random allocation of treatment to study lesions per tooth pair.
Units Other Than Participants: Lesions
Groups:
- Participants With Paired Lesions: Resin Infiltration / Control: Within-person study: both arms were applied in same participant (2 study teeth/lesions per person).
  Resin infiltration (test) or Sham Treatment (control) of two paired carious lesions in addition to preventative measures and behavioral modification.
Period: Overall Study
Arm/Group | Participants With Paired Lesions: Resin Infiltration / Control
Started | 42; 84 Lesions
Completed | 29; 58 Lesions
Not Completed | 13; 26 Lesions
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Analysis populations are single and paired lesions
Units Other Than Participants: Lesions
Groups:
- Participants With Paired Lesions: Resin Infiltration / Control: Within-person study: both arms were applied in same participant (2 study teeth/lesions per person).
Arm/Group | Participants With Paired Lesions: Resin Infiltration / Control
Number analyzed (Participants) | 42
Number analyzed (Lesions) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 11
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Number of Lesions with Progression [Count of Units; unit: Lesions] — Lesion progression is measured by assessment of single radiographs (using depth categories) and pairwise comparison of radiographs over time (continuous progression)
  Lesions | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With Progression as Measured by Pairwise (PW) Comparison (N=Lesions)
Description: Cumulative lesion progression as measured by PW comparison of radiographs (baseline versus 3 year)
Time Frame: 3 Years
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Resin Infiltration: Resin infiltration of lesion in addition to preventative measures (oral hygiene, diet counseling, repeated fluoride varnish)
- Control: Sham treatment of lesion in addition to preventative measures (oral hygiene, diet counseling, repeated fluoride varnish)
Arm/Group | Resin Infiltration | Control
Number analyzed (Participants) | 29 | 29
Number analyzed (Lesions) | 29 | 29
Lesions | 4 | 14
Statistical Analysis 1: Comparison: Resin Infiltration vs Control; Test type: Superiority; p = 0.003, McNemar

2. Secondary Outcome: Number of Lesions With Progression as Measured by Depth Category (N=Lesions)
Description: Radiographic lesion depth categories: E2 (inner enamel), D1 (outer dentin) and D2-rest (middle dentin or restored). Lesion depth assessment on single radiograph (baseline, 3 yr).
Time Frame: 3 Years
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Resin Infiltration | Control
Number analyzed (Participants) | 29 | 29
Number analyzed (Lesions) | 29 | 29
Lesions | 3 | 7
Statistical Analysis 1: Comparison: Resin Infiltration vs Control; Test type: Superiority; p = 0.17, McNemar

ADVERSE EVENTS:
Time Frame: Baseline through 3 years
Arm/Group | Participants With Paired Lesions: Resin Infiltration / Control
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT01584024/Prot_SAP_000.pdf